CLINICAL TRIAL: NCT02015039
Title: Pilot Trial of Botulinum Toxin and Occupational Therapy for Writer's Cramp
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140030; 14-N-0030
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02-13

CONDITIONS: Dystonia
Keywords: Occupational Therapy; Botulinum Toxin; Writer's Cramp
MeSH Terms: conditions — Dystonia; Dystonic Disorders | interventions — Occupational Therapy

ARMS (2):
- Botulinum Toxin Therapy Only (Active Comparator)
  Interventions: Drug: BoNT Injections
- Botulinum Toxin Therapy plus Occupational Therapy (Experimental): Intervention
  Interventions: Drug: BoNT Injections; Procedure: Occupational Therapy

INTERVENTIONS:
Drug: BoNT Injections
Procedure: Occupational Therapy
  Arms: Botulinum Toxin Therapy plus Occupational Therapy

SUMMARY:
Objective: Writer s cramp (WC) is a form of focal hand dystonia (FHD). Focal injections of botulinum toxin (BoNT) are the current best therapy. Past studies showed that some types of rehabilitative therapy can be useful. The hypothesis of this study is that BoNT together with a specific type of occupational therapy will be better than BoNT alone for treating these patients. Additionally, studies on WC were hampered by the lack of objective, validated rating scales. In this pilot study, we will assess the value of a new scale compared with older scales.

Study population: The study population will consist of 12 WC patients (accrual ceiling of 16).

Design: Patients will be randomized so that 6 patients will receive just BoNT therapy and 6 patients will receive BoNT therapy plus occupational therapy. The physical therapy will involve specific exercises of finger movements in the direction opposite to the patient s own dystonic movements, during the writing task. The movements will be isometric against splints made to suit the individual patient. The final outcome will be assessed after 20 weeks of treatment. Patients will be evaluated on several scales, including the writer s cramp rating scale (WCRS) and writer s cramp impairment scale (WCIS), and will also be videotaped. The primary outcome will be based on patient reported subjective scale and the secondary outcomes will be assessed by four blinded raters of the videotapes, done both before and after treatment.

Outcome measures: The primary outcome is to show additional improvement from baseline with BoNT therapy plus occupational therapy compared to BoNT alone at 20 weeks using a patient-rated subjective scale. The secondary outcomes are to show improvement in scores of WCRS, WCIS, WCDS, and writing parameters with a new handwriting analysis program. Additionally, the scores obtained from WCRS and WCIS will be compared.

DETAILED DESCRIPTION:
Objective: Writer s cramp (WC) is a form of focal hand dystonia (FHD). Focal injections of botulinum toxin (BoNT) are the current best therapy. Past studies showed that some types of rehabilitative therapy can be useful. The hypothesis of this study is that BoNT together with a specific type of occupational therapy will be better than BoNT alone for treating these patients. Additionally, studies on WC were hampered by the lack of objective, validated rating scales. In this pilot study, we will assess the value of a new scale compared with older scales.

Study population: The study population will consist of 12 WC patients (accrual ceiling of 16).

Design: Patients will be randomized so that 6 patients will receive just BoNT therapy and 6 patients will receive BoNT therapy plus occupational therapy. The physical therapy will involve specific exercises of finger movements in the direction opposite to the patient s own dystonic movements, during the writing task. The movements will be isometric against splints made to suit the individual patient. The final outcome will be assessed after 20 weeks of treatment. Patients will be evaluated on several scales, including the writer s cramp rating scale (WCRS) and writer s cramp impairment scale (WCIS), and will also be videotaped. The primary outcome will be based on patient reported subjective scale and the secondary outcomes will be assessed by four blinded raters of the videotapes, done both before and after treatment.

Outcome measures: The primary outcome is to show additional improvement from baseline with BoNT therapy plus occupational therapy compared to BoNT alone at 20 weeks using a patient-rated subjective scale. The secondary outcomes are to show improvement in scores of WCRS, WCIS, WCDS, and writing parameters with a new handwriting analysis program. Additionally, the scores obtained from WCRS and WCIS will be compared.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. be at least 18 years of age
  2. have writer s cramp
  3. patients are enrolled in 93-N-0202 and 85-N-0195
  4. willing to be videotaped while writing
  5. have normal hand function other than FHD
  6. be willing to use therapeutic daily rehabilitative therapies as prescribed
  7. have some positive subjective response to BoNT demonstrated on at least two prior treatments
  8. be able to comprehend and perform the daily activities required for those who are involved in combined therapy.

EXCLUSION CRITERIA

1. BoNT administration within 3 months of participation
2. No response to BoNT
3. Unable to provide consent
4. Patients taking oral medications for WC including muscle relaxants or other centrally-active medications such as antidepressants which may enhance tremors
5. Medical conditions that affect hand function, such as stroke, nerve entrapment, tremor, parkinsonism, chorea, ataxia affecting the dominant hand
6. Unable to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-12-03; Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zeuner KE, Bara-Jimenez W, Noguchi PS, Goldstein SR, Dambrosia JM, Hallett M. Sensory training for patients with focal hand dystonia. Ann Neurol. 2002 May;51(5):593-8. doi: 10.1002/ana.10174. PMID 12112105
- [Background] Zeuner KE, Hallett M. Sensory training as treatment for focal hand dystonia: a 1-year follow-up. Mov Disord. 2003 Sep;18(9):1044-7. doi: 10.1002/mds.10490. PMID 14502673
- [Background] Zeuner KE, Shill HA, Sohn YH, Molloy FM, Thornton BC, Dambrosia JM, Hallett M. Motor training as treatment in focal hand dystonia. Mov Disord. 2005 Mar;20(3):335-41. doi: 10.1002/mds.20314. PMID 15486996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with Writer's Cramp were recruited from a monthly botulinum clinic at NIH.
Pre-assignment Details: Subjects with Writer's Cramp with varying degrees of severity were randomized to receive either botulinum toxin therapy only or botulinum toxin therapy plus occupational therapy.
Groups:
- Botulinum Toxin Therapy Only: Patients with writer's cramp receive botulinum toxin therapy only. Patients in this group will be seen for 9 visits during a 24 week period, following their botulinum toxin injection. Visits 1-4 will be 1 week apart and visits 5-9 will be 4 weeks apart. Visits will entail hand grip assessment, video recording, and patient rated subjective severity scales.
- Botulinum Toxin Therapy Plus Occupational Therapy: Patients with writer's cramp receive botulinum toxin therapy plus occupational therapy. Patients in this group receive botulinum toxin injections and 10 minutes of daily writing. This group will be seen for 9 visits during a 24 week period, following their botulinum toxin injection and occupational therapy instruction. Visits 1-4 will be 1 week apart and visits 5-9 will be 4 weeks apart. Visits will entail hand grip assessment, video recording, and patient rated subjective severity scales.
Period: Overall Study
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Not eligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 62.33 [52 to 74] | 63.5 [57 to 72] | 62.92 [52 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Using a Patient Rated Subjective Scale (Visual Analogue Scale), Change From Baseline With Botulinum Toxin Therapy Plus Occupational Therapy Compared to Botulinum Toxin Therapy Alone at 20 Weeks.
Description: A visual analogue scale was used to rate patient's subjective rating of the severity of their writer's cramp at each visit. Patients were asked to mark the location on a 10 centimeter line corresponding to the severity of their writer's cramp. Ratings ranged from "mild" disease severity to "severe" disease severity. The mark was measured on the 10 centimeter line, ranging from 0 to 10. The percent change in the patient rated subject scale was measured at baseline (Visit 1) and 20 weeks (Visit 8) in the two groups.
Time Frame: Baseline and 20 weeks
Population: The patient rated subjective scale was not administered at baseline in two subjects, i.e., one subject in each group, therefore these subjects were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 5 | 5
percentage of change | -20.6 (49.3) | -41.6 (36.5)

2. Secondary Outcome: Change in the Writers Cramp Rating Scale (WCRS) From Baseline to Week 20 in Participants Receiving Botulinum Toxin Therapy Alone Compared With Botulinum Toxin Therapy Plus Occupational Therapy.
Description: The Writers Cramp Rating Scale (WCRS) is a tool used to quantify the treatment effect of local botulinum toxin injections in writer's cramp using writing performance and a computer assisted analysis of writing speed. The WCRS consists of two parts. Part A provides a writing movement score measuring 1) dystonic posture elbow score (ES: 0-2), 2) wrist score (WRS: 0-4), 3) finger score (FS: 0-6), 4) latency of dystonia (L: 1-2) and 5) writing tremor (WT: 0-2). The writing movement sub-score is calculated as (ES + WRS + FS) x L + (WT x 2) (0-28). Part B provides an assessment of writing speed (WS: 0-2). The WCRS score is the total of the writing movement sub-score and the writing speed sub-score. The total WCRS range is between "0" indicating absent residual writer's cramp symptoms to "30" indicating severe writer's cramp symptoms. The percentage change in the WCRS was measured at baseline (Visit 1) and 20 weeks (Visit 8) in the two groups.
Time Frame: Baseline and 20 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 6 | 6
percentage of change | 46 (37.2) | -20.18 (37.0)

3. Secondary Outcome: Change on the Writer's Cramp Impairment Scale (WCIS) Score From Baseline to 20 Weeks.
Description: The Writer's Cramp Impairment Scale (WCIS) scale assesses the speed of writing, the number of breaks during writing, the occurrence and intensity of involuntary (pathological) postures/abnormal movements (while writing, while performing repetitive wrist movements), the degree of tremor that occurs while performing repetitive spiral movements, and the presence of mirror movements. The scale ranges from 0-180 with 0 representing "no impairment" and 180 representing "severe impairment". The percent change in the WCIS was measured at baseline (Visit 1) and 20 weeks (Visit 8) in the two groups.
Time Frame: Baseline and 20 weeks
Population: The Writer's Cramp Impairment Scale (WCIS) was not collected at week 20 for two subjects in the Botulinum Toxin Therapy plus Occupational Therapy group, therefore these two subjects were not included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 6 | 4
percentage of change | 7.61 (9.9) | -34.13 (31.77)

4. Secondary Outcome: Change on the Writer's Cramp Disability Scale (WCDS) Score From Baseline to 20 Weeks.
Description: The Writer's Cramp Disability Scale (WCDS) is a self-reported questionnaire which queries patients regarding problems they experience with writing and other every day activities due to writer's cramp. The scale ranges from 0-42 with 0 representing "no difficulty" and 42 representing "marked difficulty". The percent change in the WCDS was measured at baseline (Visit 1) and 20 weeks (Visit 8) in the two groups.
Time Frame: Baseline and 20 weeks
Population: The Writer's Cramp Disability Scale (WCDS) was not administered at baseline for one subject in the Botulinum Toxin Therapy Only group therefore this subject was not included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 5 | 6
percentage of change | -41.5 (26.00) | -35.6 (11.44)

5. Secondary Outcome: Change in Hand Grip Strength From Baseline to 20 Weeks Following Botulinum Toxin Therapy Alone and Botulinum Toxin Therapy Plus Occupational Therapy.
Description: Hand grip strength was measured using a commercially available dynamometer. The dynamometer instrument measures maximum isometric strength of the hand and forearm muscles. Hand grip strength was measured with the dynamometer during each visit. The percent change in hand grip strength between baseline (Visit 1) and 20 weeks (Visit 8) in the two groups.
Time Frame: Baseline and 20 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 6 | 6
percentage of change | 7.49 (46.9) | -9.00 (25.9)

6. Secondary Outcome: Change in Quantitative Writing Metrics Obtained Via Numerical Analyses of Writing Samples Using a Digitizing Tablet.
Description: Subjects with writer's cramp were instructed to draw with their dominant hand between the lines of a 5-loop Archimedes spiral presented on a paper placed over the surface of a digitizing tablet sampling pen tip position at a 100 Hz. The deviation of the drawn spiral to the ideal spiral was calculated at each sampled point. The root mean square of the total spiral error was used as a measure of dysfunctional pen control in subjects with writer's cramp compared with normative data. The percent change of the root mean square was calculated at baseline (Visit 1) and 20 weeks (Visit 8) in the two groups.
Time Frame: Baseline and 20 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 6 | 6
percentage of change | 25.76 (54.17) | -0.91 (21.98)

7. Secondary Outcome: Using a Patient Rated Subjective Scale (Visual Analogue Scale), Change From Baseline With Botulinum Toxin Therapy Plus Occupational Therapy Compared to Botulinum Toxin Therapy Alone at 24 Weeks.
Description: A visual analogue scale was used to rate patient's subjective rating of the severity of their writer's cramp at each visit. Patients were asked to mark the location on a 10 centimeter line corresponding to the severity of their writer's cramp. Ratings ranged from "mild" disease severity to "severe" disease severity. The mark was measured on the 10 centimeter line, ranging from 0 to 10. The percent change in the patient rated subject scale was measured at baseline (Visit 1) and 24 weeks (Visit 9) in the two groups.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
Number analyzed (Participants) | 5 | 5
percentage of change | -2.12 (74.7) | -2.0 (69.6)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Botulinum Toxin Therapy Only | Botulinum Toxin Therapy Plus Occupational Therapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes